CLINICAL TRIAL: NCT04808791
Title: A Study to Evaluate the Safety and Feasibility of Irinotecan, Trifluridine/Tipiracil (TAS-102), and Oxaliplatin (iTTo) for Treatment Naive Advanced Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma
Brief Title: iTTo for Treatment Naive Advanced Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-0022
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Gastroesophageal Junction Adenocarcinoma; Advanced Gastric Carcinoma
MeSH Terms: interventions — Irinotecan; Oxaliplatin; trifluridine tipiracil drug combination; Trifluridine; tipiracil

STUDY DESIGN:
Intervention Model Description: A single arm, interventional study combining Irinotecan, Trifluridine/Tipiracil (TAS-102), and Oxaliplatin (iTTo)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm iTTO treatment (Experimental): Patients will receive the combination of irinotecan, TAS-102, and Oxaliplatin on a 28 day cycle with the following doses;
  * Irinotecan 160mg/m2 IV infusion over 60-90 mins on day 1
  * Oxaliplatin 100mg/m2 IV infusion over 2 hours on day 1
  * TAS-102 (Trifluridine/Tipiracil) 25mg/m2 twice a day, on days 1-5 and 8-12 every 28days.
  Interventions: Drug: Irinotecan; Drug: Oxaliplatin; Drug: TAS 102 (Trifluridine/Tipiracil)

INTERVENTIONS:
Drug: Irinotecan — Irinotecan is an anti-cancer ("antineoplastic" or "cytotoxic") chemotherapy drug. This medication is classified as a "plant alkaloid" and "topoisomerase I inhibitor."
  Other Names: Camptosar
Drug: Oxaliplatin — Oxaliplatin is an anti-cancer ("antineoplastic" or "cytotoxic") chemotherapy drug. Oxaliplatin is classified as an "alkylating agent."
  Other Names: Eloxatin
Drug: TAS 102 (Trifluridine/Tipiracil) — Trifluridine/Tipiracil is an anti-cancer ("antineoplastic" or "cytotoxic") chemotherapy drug. This medication is classified as an antimetabolite/pyrimidine analog; antimetabolite/thymidine phosphorylase inhibitor
  Other Names: Lonsurf

SUMMARY:
This study will evaluate the safety and feasibility of Irinotecan, Trifluridine/Tipiracil (TAS-102) and Oxaliplatin (iTTo) for treatment naïve advanced gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age or older.
2. Histologically documented locally advanced or metastatic gastric or GEJ adenocarcinoma not previously treated with palliative systemic therapy.
3. Patients must be capable of providing consent to enrolment and treatment.
4. Patients with a performance status of ECOG 0-1 will be eligible for enrolment (see appendix 1).
5. Measurable disease must be present according to RECIST criteria V1.1 (see appendix ).
6. Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test at the time of screening. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy or bilateral salpingectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes.
7. Patients (men and women) of childbearing / reproductive potential should use highly effective birth control methods, as defined by the investigator, during the study treatment period and for a period of 6 months after the last dose of study drug. A highly effective method of birth control is defined as those that result in low failure rate (i.e. less than 1% per year) when used consistently and correctly. Note: abstinence is acceptable if this is established and preferred contraception for the patient and is accepted as a local standard.
8. Female patients who are breast-feeding should discontinue nursing prior to the first dose of study treatment and until 30 days after the last dose of study drug.
9. Male patients should agree to not donate sperm during the study and for a period of at least 6 months after last dose of study drug.
10. Absence of any condition hampering compliance with the study protocol and follow- up schedule; those conditions should be discussed with the patient before registration in the trial.
11. Patients may have received prior surgery if this surgery was ≥ 4 weeks before study entry and patients must have recovered from the toxic effects of this treatment.
12. Patients who have treated brain metastasis (via local radiation standards or surgical resection or local ablative techniques) and who are either off steroids or on a stable dose of steroids for at least one month (30 days), AND who are off anticonvulsants, AND have radiological documented stability of lesions for at least 3 months may be eligible. Each case should be discussed with the study Chair.
13. Patients who have received prior chemotherapy or radiation delivered as part of initial curative therapy (i.e. neoadjuvant or adjuvant chemotherapy administered alone and/or concurrently delivered with radiation and/or surgery) are permitted as long as that treatment was completed at least 6 months prior to study start date.
14. Patients may have received prior palliative radiotherapy (unless radiation was curative therapy to pelvis or to ≥ 25% of bone marrow stores) if this radiation was ≥ 4 weeks before study entry and patients must have recovered from the toxic effects of this treatment.
15. Patients with unknown Her2/neu status, or negative Her2/neu status based on IHC and/or FISH/CISH (Testing does not need to be done unless it is standard of care at participating centres).
16. The following adequate organ function laboratory values must be met:

Hematological:

Absolute neutrophil count (ANC) >1.5 x10^9/L Platelet count >100 x10^9/L Hemoglobin >8 g/dL (may have been transfused)

Renal:

serum creatinine ≤ upper limit of institutional normal OR calculated creatinine clearance of ≥ 50 mL/min using the Cockcroft-Gault formula (or local institutional standard method)

Hepatic:

Total serum bilirubin <1.5x ULN AST and ALT <2.5x ULN (or ≤ 5 x ULN for patients with documented metastatic disease to the liver)

Exclusion Criteria:

1. Patients who have received prior palliative chemotherapy for their advanced gastric or GEJ tumor.
2. Prior curative or palliative radiation treatment to the pelvis or radiation therapy to ≥ 25% of bone marrow stores.
3. History of bowel obstruction due to peritoneal metastases or clinically documented ascites requiring paracenteses.
4. Previous or concurrent malignancies, excluding curatively treated in situ carcinoma of the cervix or uterus or non-melanoma skin cancer or in-situ carcinoma of the prostate (Gleason score ≤ 7, with all treatment being completed 6 months prior to enrollment, unless at least 5 years have elapsed since last treatment and the patient is considered cured).
5. Active bacterial, viral, or fungal infection(s) requiring systemic therapy, defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment.
6. Known infection with hepatitis B or C, or history of human immunodeficiency virus (HIV) infection, or subject receiving immunosuppressive or myelosuppressive medications that would, in the opinion of the investigator, increase the risk of serious neutropenic complications.
7. Any serious medical condition within 6 months prior to study entry such as myocardial infarction, uncontrolled congestive heart failure, unstable angina, active cardiomyopathy, unstable ventricular arrhythmia, cerebrovascular diseases, uncontrolled hypertension, uncontrolled diabetes, uncontrolled psychiatric disorder, serious infection, active peptic ulcer disease, or other medical condition that may be aggravated by treatment.
8. Pre-existing neuropathy ≥ grade 2 from any cause.
9. Patients with unstable metastasis to the central nervous system (CNS). A CT scan or MRI is NOT required to rule out brain metastases unless there is clinical suspicion of CNS involvement.
10. Pregnant or lactating women; women of child bearing potential must have a negative serum pregnancy test within 7 days of trial registration. Women or men of child bearing potential must use effective contraception (defined by the treating physician) which must be documented in study CRFs.
11. History of allergic reaction to planned study medications.
12. Patient has a ≥ 20% decrease in serum albumin level between baseline visit, if available, and within 72 hours prior to first study treatment dose.
13. Patient is on coumadin.
14. History of interstitial lung disease.
15. History of connective tissue disorders (e.g. lupus, scleroderma, polyarteritis nodosa).
16. Enrollment in any other clinical protocol or investigational study with an interventional agent or assessments that may interfere with study procedures.
17. Any significant medical condition, laboratory abnormality, or psychiatric illness, that would prevent the subject from participating in the study, places the subject at unacceptable risk if he/she were to participate in the study, or any condition that confounds the ability to interpret data from the study.
18. Positive Her2/neu status (NOTE: if this is discovered after patient has already been enrolled on study, patient may continue on study per the discretion of the treating physician.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
The number of participants who complete at least 2 cycles of iTTo for the treatment of advanced gastric and GEJ cancers, over the total duration of study | 1 year after enrolment of last participant.
  The number of participants who complete at least 2 cycles of iTTo for the treatment of advanced gastric and GEJ cancers, over the total duration of study.
Safety/Tolerability | Through study completion, up to 2 years.
  Treatment related and non-related adverse events per CTCAE v.5.0 of iTTo for the treatment of advanced gastric and GEJ cancers. Incidence of adverse events, the number of dose modifications and discontinuations due to adverse events.

SECONDARY OUTCOMES:
Objective Response Rate | 1 year after enrollment of last participant.
  Defined as the proportion of participants achieving either a partial response or a complete response as best-overall response per RECIST criteria 1.1
Progression Free Survival | 5 years from final study drug dose.
  Defined as the time between the date of treatment initiation and the date of disease progression or death.
Overall Survival | 5 years from final study drug dose.
  Defined as the time between the date of treatment initiation and the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Hatim Karachiwala, MD, Principal Investigator — Alberta Health Services - Cross Cancer Institute
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada